CLINICAL TRIAL: NCT05682729
Title: The Early Development of Flexible Attention to Numerical and Spatial Magnitudes: Clinical Trial
Brief Title: Flexible Attention to Magnitudes and Early Math
Acronym: FAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Dayton (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: R15HD100936 (NIH)
Record Dates: First submitted 2022-12-19; First posted 2023-01-12 (Actual); Results first posted 2025-10-30 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Mathematics Abilities

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Size to Number (Experimental)
  Interventions: Behavioral: Book Reading Intervention
- Mixed (Experimental)
  Interventions: Behavioral: Book Reading Intervention
- Traditional Counting (Active Comparator)
  Interventions: Behavioral: Book Reading Intervention
- Non-Numerical Control (Placebo Comparator)
  Interventions: Behavioral: Book Reading Intervention

INTERVENTIONS:
Behavioral: Book Reading Intervention — Children read books containing relevant stimuli.

SUMMARY:
The goal of this clinical trial is to test the malleability of preschool-aged children's flexible attention to numerical and spatial magnitudes. The main questions it aims to answer are: Does a flexible attention to magnitudes intervention improve young children's math abilities in the area of flexible attention to magnitudes as well as executive functioning and number line estimation skills? Does this intervention improve young children's math abilities more than a traditional counting intervention? "Does the method of flexible attention to magnitudes intervention affect how much children improve in their math abilities?

Participants will complete a pre-test and post-test in their math abilities and three intervention sessions with a trained experimenter. Each intervention session will involve reading researcher-created books with one-on-one with children for about 20 minutes. Children will be assigned to one of four intervention conditions:

* Size to Number Intervention Condition
* Size and Number Mixed Intervention Condition
* Traditional Counting Intervention
* Non-Numerical Control Intervention

DETAILED DESCRIPTION:
This experiment will test the following hypothesis: Children's flexible attention to magnitudes (FAM) ability is malleable and can be developed through innovative interventions. The experiment will include a clinical trial to assess the feasibility of a future clinical intervention to improve children's FAM ability for children at-risk for math difficulties.

Participants. Using results from recent number book interventions (ηp2 = .094; Gibson, Gunderson, & Levine, under review), an estimated sample size of 116 preschool-aged children (3 - 5 years old), or 29 children per group, will be recruited. An additional 8 participants will be recruited to account for any possible attrition during the course of the experiment.

Method and Analyses. Children will be randomly assigned to one of 4 conditions: Size to Number condition, Mixed condition, or one of two control conditions - a Traditional Counting condition or an Non-Numerical Control condition. In each condition, children will complete a pre-test, followed by three intervention sessions with an experimenter, then a post-test. All assessments and intervention sessions will be completed in a one-on-one setting with an experimenter in a quiet area of the child's childcare center or school. Each condition will involve playing a game on a tablet with an experimenter, and the premise of each game will be children going to the zoo. All stimuli for conditions will be created by the University of Dayton computer engineering students in their research and design course. The stimuli for the Size to Number and Mixed conditions will be identical where all trials are incongruent with respect to numerical and spatial magnitudes across sets, but the ordering of instructions and item presentation will differ. In the Size to Number condition, children will view two sets of animals, each enclosed by a box, and will be asked to indicate which set has bigger animals. Children will then switch to a condition in which they are asked to switch and indicate which set has more animals, with 10 trials for both the number and size conditions. Children will receive feedback on each trial. In the Mixed condition, children will receive 20 trials in which size and number trials are intermixed. In the Traditional Counting condition, children will only see congruent numerical and spatial magnitudes, in other words, sets where the object set with more items will also have larger items and the set with fewer items will also have smaller items. Children will be asked to compare these sets, and feedback will be given. Finally, in the Non-Numerical Control condition, children will see various animals on each trial and will be asked to give the animal's name and sound.

An ANCOVA will be used to analyze participant data, with the 4 conditions as the between-subjects variable, and covariates will include children's pre-test, age, gender, and language. The investigator expects to find that both the Size to Number and Mixed conditions will produce higher FAM post-test scores compared to the Traditional Counting and Non-Numerical Control conditions, but do not have a specific prediction as to whether or not the Size to Number or Mixed conditions will outperform one another. The assessments administered at pre- and post-test will include the FAM task, and the investigator will also explore possible transfer effects to children's executive functioning skills and their number line estimation abilities.

ELIGIBILITY:
Inclusion Criteria:

* Child ages 3 - 5

Exclusion Criteria:

-

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 116 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Early Childhood Education Facilities, Dayton, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Anonymized pre- and post-test scores will be shared.
Supporting Information: Study Protocol
Time Frame: Data available when published through the Open Science Framework (OSF).

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: We initially recruited 169 participants for the study, knowing that school absences during a short-term weeklong study would likely significantly reduce the final sample size. Participant exclusions were primarily due to school absences (n = 28), children not wanting to participate in one or more assessments (n = 13), developmental delays (n = 1), and technical errors with the online data collection system (n = 11).
Period: Overall Study
Arm/Group | Size to Number | Mixed | Traditional Counting | Non-Numerical Control
Started | 37 | 25 | 30 | 24
Completed | 37 | 25 | 30 | 24
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The population for analysis is the same as in participant flow.
Groups:
- Total: Total of all reporting groups
Arm/Group | Size to Number | Mixed | Traditional Counting | Non-Numerical Control | Total
Number analyzed (Participants) | 37 | 25 | 30 | 24 | 116
Age, Continuous [Mean (Standard Deviation); unit: Months of age] | 55 (8) | 55 (8) | 56 (8) | 56 (8) | 56 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 14 | 16 | 16 | 63
  Male | 20 | 11 | 14 | 8 | 53
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 4 | 5 | 10
  Not Hispanic or Latino | 31 | 21 | 23 | 17 | 92
  Unknown or Not Reported | 5 | 4 | 3 | 2 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 10 | 9 | 5 | 8 | 32
  White | 18 | 9 | 14 | 7 | 48
  More than one race | 3 | 3 | 5 | 7 | 18
  Unknown or Not Reported | 6 | 4 | 6 | 2 | 18
Region of Enrollment [Number; unit: participants]
  United States | 37 | 25 | 30 | 24 | 116

OUTCOME MEASURES:

1. Primary Outcome: Change in Flexible Attention to Magnitudes Task
Description: Assesses preschool-aged children's ability to flexibly shift between attending to numerical and spatial magnitudes. The task is scored for accuracy (0 - 1), and higher scores indicate better outcomes. The outcome measure was change in accuracy from baseline to immediately after intervention, or 4 days.
Time Frame: Baseline and after intervention (up to 4 days)
Population: The population was children who completed baseline and post-intervention assessment.
Measure: Mean (Standard Deviation); unit: mean pre-post diff in units on a scale
Groups:
- Size to Number: Children read books that contained questions about spatial magnitude comparisons followed by questions about numerical magnitude comparisons.
- Mixed: Children read books that contained questions about spatial and numerical magnitude comparisons that were intermixed throughout the books.
- Traditional Counting: Children read books that focused on counting.
- Non-Numerical Control: Children read books with questions about shapes and colors.
Arm/Group | Size to Number | Mixed | Traditional Counting | Non-Numerical Control
Number analyzed (Participants) | 37 | 25 | 30 | 24
mean pre-post diff in units on a scale | .07 (.17) | .13 (.23) | .03 (.26) | .08 (.23)
Statistical Analysis 1: Comparison: Size to Number vs Mixed vs Traditional Counting vs Non-Numerical Control; We specifically compared the pre-to-post test change in accuracy on the FAM task across the four groups using a within-subjects ANCOVA and specifically a group by time (pre-to-post test) interaction. We controlled for age, gender, and children's executive function skills; Test type: Superiority; p = .41, ANCOVA — A priori threshold for statistical significance was p < .05. Wilks' Lambda F(3, 109) = .96, p = .41, ηp2 = .03; Partial Eta Squared = .03
Statistical Analysis 2: Comparison: Mixed; Following the omnibus test, we conducted planned comparisons to compare pre-to-post test change within our experimental and control groups to test for significant positive change from pre-to-post test; Test type: Superiority; p = .004, ANCOVA; Partial Eta Squared = .07
Statistical Analysis 3: Comparison: Size to Number; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = .031, ANCOVA; Partial Eta Squared = .04
Statistical Analysis 4: Comparison: Traditional Counting; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = .463, ANCOVA; Partial Eta Squared = .01
Statistical Analysis 5: Comparison: Non-Numerical Control; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = .186, ANCOVA; Partial Eta Squared = .02

2. Secondary Outcome: Change in Minnesota Executive Function Scale
Description: Ipad based card game assessing attention shifting. Standardized scores are calculated, with a mean of 100 and a standard deviation of 15. The mean change in standard score from pre-to-post test was examined across all 4 groups.
Time Frame: baseline and immediately after intervention (up to 4 days)
Population: The population was children who completed baseline and post-intervention assessment.
Measure: Mean (Standard Deviation); unit: mean pre-post diff on score on a scale
Groups:
- Size to Number: Children read books containing questions about spatial numerical magnitudes followed by numerical magnitude comparisons.
- Mixed: Children read books containing intermixed spatial and numerical magnitude comparison questions.
- Counting: Children read books about counting.
- Non-Numerical Control: Children read books about shapes and colors.
Arm/Group | Size to Number | Mixed | Counting | Non-Numerical Control
Number analyzed (Participants) | 37 | 25 | 30 | 24
mean pre-post diff on score on a scale | -.51 (7.36) | 1.12 (5.19) | -1.2 (10.21) | 3.96 (7.36)
Statistical Analysis 1: Comparison: Size to Number vs Mixed vs Counting vs Non-Numerical Control; Test type: Superiority; p = .605, ANCOVA; Partial Eta Squared = .02

3. Secondary Outcome: Change in Number Line Estimation Task
Description: Child identifies location of a number on a 0 - 10 number line. Total scores range from 0 - 20, with higher scores indicating better performance. Pre-to-post test change scores were examined.
Time Frame: baseline and immediately after (up to 4 days)
Population: The population was children who completed baseline and post-intervention assessment.
Measure: Mean (Standard Deviation); unit: Mean pre-post diff on score on a scale
Groups:
- Size to Number: Children read books that included questions about spatial magnitude comparisons followed by questions about numerical magnitude comparisons.
- Mixed: Children read books that contained intermixed questions about spatial and numerical magnitude comparisons.
Arm/Group | Size to Number | Mixed | Counting | Non-Numerical Control
Number analyzed (Participants) | 37 | 25 | 30 | 24
Mean pre-post diff on score on a scale | .51 (1.68) | .32 (1.49) | -.17 (1.78) | -.38 (1.53)
Statistical Analysis 1: Comparison: Size to Number vs Mixed vs Counting vs Non-Numerical Control; Test type: Superiority; p = .618, ANCOVA; Partial Eta Squared = .02

ADVERSE EVENTS:
Time Frame: 4 days
Arm/Group | Size to Number | Mixed | Traditional Counting | Non-Numerical Control
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/25 | 0/30 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/25 | 0/30 | 0/24
Other Adverse Events (participants affected / at risk) | 0/37 | 0/25 | 0/30 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-06-30): https://cdn.clinicaltrials.gov/large-docs/29/NCT05682729/Prot_SAP_000.pdf